CLINICAL TRIAL: NCT02128490
Title: A Phase 2, Randomized, Double Blind, Multicenter, Placebo Controlled Study to Evaluate the Efficacy and Safety of Febuxostat 40 mg XR, 80 mg XR, 40 mg IR and 80 mg IR in Subjects With Gout and Moderate Renal Impairment
Brief Title: Efficacy and Safety of Extended Release and Immediate Release Febuxostat in Participants With Gout and Moderate Renal Impairment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FEB-XR_201; U1111-1152-3942 (Other: World Health Organization)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-09

CONDITIONS: Gout; Moderate Renal Impairment
Keywords: Drug therapy
MeSH Terms: conditions — Gout | interventions — Febuxostat; Colchicine; Naproxen; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Febuxostat IR 40 mg (Active Comparator): Febuxostat Immediate Release (IR) 40 mg over-encapsulated tablet, orally, once daily, and colchicine 0.6 mg tablet, orally, every other day, or, naproxen 250 mg tablets, orally, twice a day and lansoprazole 15 mg capsule, orally once daily, for 3 months.
  Interventions: Drug: Febuxostat IR; Drug: Colchicine; Drug: Naproxen; Drug: Lansoprazole
- Febuxostat IR 80 mg (Active Comparator): Febuxostat IR 80 mg over-encapsulated tablet, orally, once daily, and colchicine 0.6 mg tablet, orally, every other day, or, naproxen 250 mg tablets, orally, twice a day and lansoprazole 15 mg capsule, orally once daily, for 3 months.
  Interventions: Drug: Febuxostat IR; Drug: Colchicine; Drug: Naproxen; Drug: Lansoprazole
- Febuxostat XR 40 mg (Experimental): Febuxostat Extended Release (XR) 40 mg over-encapsulated capsule, orally, once daily, and colchicine 0.6 mg tablet, orally, every other day, or, naproxen 250 mg tablets, orally, twice a day and lansoprazole 15 mg capsule, orally once daily, for 3 months.
  Interventions: Drug: Febuxostat XR; Drug: Colchicine; Drug: Naproxen; Drug: Lansoprazole
- Febuxostat XR 80 mg (Experimental): Febuxostat XR 80 mg over-encapsulated capsule, orally, once daily, and colchicine 0.6 mg tablet, orally, every other day, or, naproxen 250 mg tablets, orally, twice a day and lansoprazole 15 mg capsule, orally once daily, for 3 months.
  Interventions: Drug: Febuxostat XR; Drug: Colchicine; Drug: Naproxen; Drug: Lansoprazole
- Placebo (Placebo Comparator): Febuxostat placebo-matching capsule, orally, once daily, and colchicine 0.6 mg tablet, orally, every other day, or, naproxen 250 mg tablets, orally, twice a day and lansoprazole 15 mg capsule, orally once daily, for 3 months.
  Interventions: Drug: Febuxostat placebo; Drug: Colchicine; Drug: Naproxen; Drug: Lansoprazole

INTERVENTIONS:
Drug: Febuxostat IR — Febuxostat IR over-encapsulated tablets
  Other Names: Uloric
  Arms: Febuxostat IR 40 mg; Febuxostat IR 80 mg
Drug: Febuxostat XR — Febuxostat over-encapsulated capsules
  Arms: Febuxostat XR 40 mg; Febuxostat XR 80 mg
Drug: Febuxostat placebo — Febuxostat IR and XR placebo-matching capsules
  Arms: Placebo
Drug: Colchicine — Colchicine tablets
Drug: Naproxen — Naproxen tablets
Drug: Lansoprazole — Lansoprazole capsules

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of febuxostat 40 mg extended release (XR) and 80 mg XR in comparison with febuxostat 40 mg immediate release (IR) and 80 mg IR, respectively, in gout participants with moderate renal impairment.

DETAILED DESCRIPTION:
The drug being tested in this study is called febuxostat. Febuxostat is being tested to decrease and maintain serum urate in people who have gout with moderate renal impairment. This study will look at serum urate levels in people who take febuxostat extended release (XR) capsules compared to febuxostat immediate release (IR) capsules and placebo.

The study will enroll approximately 200 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the five treatment groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Febuxostat 40 mg XR
* Febuxostat 80 mg XR
* Febuxostat 40 mg IR
* Febuxostat 80 mg IR
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient.

All participants will be asked to take one capsule at the same time each day throughout the study, and will be asked to call an interactive voice response system any time they are having a gout flare up. In addition to study medication, participants will also take 0.6 mg of colchicine every other day or naproxen 250 mg twice a day with lansoprazole 15 mg once a day to prevent gout flare ups.

This multi-center trial will be conducted in the United States. The overall time to participate in this study is up to approximately 4 months and participants will make up to 7 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedure.
3. Has a history or presence of gout defined as having one or more of the American Rheumatism Association (ARA) criteria for the diagnosis of gout:

   1. A tophus proven to contain urate crystals by chemical or polarized light microscopic means, AND/OR;
   2. Characteristic urate crystals in the joint fluid, AND/OR;
   3. History of at least 6 of the following clinical, laboratory, and x-ray phenomena:

   i. more than one attack of acute arthritis, ii. maximum inflammation developed within 1 day, iii. monoarticular arthritis, iv. redness observed over joints, v. first metatarsophalangeal joint painful or swollen, vi. unilateral first metatarsophalangeal joint attack, vii. unilateral tarsal joint attack, viii. tophus (proven or suspected), ix. Hyperuricemia, x. asymmetric swelling within a joint on x-ray, xi. subcortical cysts without erosions on x-ray, xii. joint fluid culture negative for organisms during attack.
4. Is male or female at least 18 years of age, inclusive.
5. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.
6. Have a serum urate (sUA) level ≥8.0 mg/dL at the Day -4 Visit or at the retest visit.
7. Has an estimated Glomerular Filtration Rate (eGRF) [Modification of Diet in Renal Disease (MDRD)] ≥30 mL/min and <60 mL/min at Screening visit (Day -21 for participants on urate lowering therapy (ULT) and Day -4 for participants not on ULT) or at the retest visit.
8. Has at least one gout flare within 12 months prior to Screening visit.

Exclusion Criteria:

1. Has received any investigational compound within 30 days prior to Screening.
2. Is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
3. Is breastfeeding or pregnant.
4. Has secondary hyperuricemia (eg, due to myeloproliferative disorder).
5. Has a history of xanthinuria.
6. Has received ULT (ie, allopurinol, probenecid, etc.) within 20 days prior to Day 1/Randomization Visit.
7. Has a known hypersensitivity to febuxostat or any components of their formulation; has a known hypersensitivity to naproxen, any other nonsteroidal anti-inflammatory drug (NSAID), aspirin, lansoprazole, colchicine or any components in their formulation.
8. Has active peptic ulcer disease.
9. Has a history of cancer (other than basal cell carcinoma of the skin) within 5 years prior to the Screening Visit.
10. Has alanine aminotransferase (ALT) and aspartate aminotransferase (AST) values >2 x the upper limit of normal (ULN).
11. Has rheumatoid arthritis which requires treatment.
12. Has a significant medical condition and/or conditions that would interfere with the treatment, safety, or compliance with the protocol.
13. Has experienced either a myocardial infarction (MI), stroke, hospitalized unstable angina, cardiac or cerebrovascular revascularization procedure or hospitalized transient ischemic attack (TIA).
14. Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 5 years prior to the Screening visit. Participant consumes >14 alcoholic beverages/week.
15. Has participated in another investigational study within the 30 days prior to the Screening Visit.
16. Has a known history of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
17. Is required to take excluded medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (89):
- United States (89):
  - Birmingham, Alabama
  - Muscle Shoals, Alabama
  - Phoenix, Arizona
  - Benny Green MD PA Family Practice, Little Rock, Arkansas
  - Little Rock, Arkansas
  - Bellflower, California
  - Escondido, California
  - Harbor City, California
  - Huntington Park, California
  - Irvine, California
  - Lomita, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Brigid Freyne MD, Murrieta, California
  - Murrieta, California
  - Orange, California
  - Rancho Cucamonga, California
  - Redondo Beach, California
  - Sacramento, California
  - San Jose, California
  - San Ramon, California
  - Clearwater, Florida
  - Coral Gables, Florida
  - Coral Springs, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Edgewater, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Miami Lakes, Florida
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Plantation, Florida
  - Port Charlotte, Florida
  - Saint Cloud, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Dunwoody, Georgia
  - East Point, Georgia
  - Suwanee, Georgia
  - East West Medical Research Institute, Honolulu, Hawaii
  - Honolulu, Hawaii
  - Brownsburg, Indiana
  - Manhattan, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Central Kentucy Reseach Associates, Lexington, Kentucky
  - Lexington, Kentucky
  - Paducah, Kentucky
  - Mandeville, Louisiana
  - Metairie, Louisiana
  - Fall River, Massachusetts
  - Detroit, Michigan
  - Kalamazoo, Michigan
  - Hazelwood, Missouri
  - Washington, Missouri
  - Las Vegas, Nevada
  - Albuquerque, New Mexico
  - Columbiana, North Carolina
  - Greensboro, North Carolina
  - Salisbury, North Carolina
  - Wilmington, North Carolina
  - Fargo, North Dakota
  - Franklin, Ohio
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Columbia, South Carolina
  - Greer, South Carolina
  - Old Point Station, South Carolina
  - Clarksville, Tennessee
  - Knoxville, Tennessee
  - Remesh C Gupta MD, Memphis, Tennessee
  - Memphis, Tennessee
  - Austin, Texas
  - Bellaire, Texas
  - 3rd Coast Research Associates, Corpus Christi, Texas
  - Corpus Christi, Texas
  - Nassau Bay, Texas
  - Plano, Texas
  - Sun Research Institute, San Antonio, Texas
  - Briggs Clinical Research LLC, San Antonio, Texas
  - San Antonio, Texas
  - Bountiful, Utah
  - Newport News, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Virginia Beach, Virginia

REFERENCES:
- [Derived] Gunawardhana L, Becker MA, Whelton A, Hunt B, Castillo M, Saag K. Efficacy and safety of febuxostat extended release and immediate release in patients with gout and moderate renal impairment: phase II placebo-controlled study. Arthritis Res Ther. 2018 May 30;20(1):99. doi: 10.1186/s13075-018-1593-0. PMID 29848361

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 65 investigative sites in the United States from 5 May 2014 to 23 October 2015.
Pre-assignment Details: Participants with a diagnosis of gout were enrolled equally in 1 of 5 treatment groups once a day: placebo, febuxostat 40 mg extended release (XR), febuxostat 80 mg XR, febuxostat 40 mg immediate release (IR) or febuxostat 80 mg IR.
Period: Overall Study
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg
Started | 38 | 37 | 39 | 37 | 38
Completed | 33 | 31 | 34 | 31 | 31
Not Completed | 5 | 6 | 5 | 6 | 7
Not completed — Pretreatment Event/Adverse Event | 1 | 0 | 1 | 1 | 0
Not completed — Major Protocol Deviation | 1 | 2 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — Voluntary Withdrawal | 3 | 3 | 1 | 1 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0 | 0
Not completed — Withdraw from Study Drug, Gout Flare | 0 | 0 | 0 | 0 | 1
Not completed — Other Miscellaneous Reasons | 0 | 0 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of double-blind study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg | Total
Number analyzed (Participants) | 38 | 37 | 39 | 37 | 38 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (12.78) | 61.3 (10.09) | 64.4 (11.21) | 63.5 (10.33) | 61.4 (12.17) | 63.1 (11.34)
Age, Customized [Number; unit: participants]
  < 45 years | 1 | 3 | 1 | 0 | 4 | 9
  45 to < 65 years | 14 | 16 | 15 | 18 | 18 | 81
  >= 65 years | 23 | 18 | 23 | 19 | 16 | 99
Age, Customized [Number; unit: participants]
  18 to < 65 years | 15 | 19 | 16 | 18 | 22 | 90
  65 to < 85 years | 21 | 18 | 23 | 19 | 16 | 97
  >= 85 years | 2 | 0 | 0 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 13 | 9 | 9 | 55
  Male | 26 | 25 | 26 | 28 | 29 | 134
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 2 | 1 | 2 | 4 | 9
  Black or African American | 4 | 10 | 10 | 12 | 10 | 46
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 2 | 0 | 4
  White | 33 | 24 | 26 | 21 | 22 | 126
  Other: Multi-racial | 0 | 1 | 1 | 0 | 2 | 4
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 2 | 1 | 7 | 7 | 7 | 24
  Not Hispanic or Latino | 36 | 36 | 32 | 30 | 31 | 165
Region of Enrollment [Number; unit: participants]
  United States | 38 | 37 | 39 | 37 | 38 | 189
Height [Mean (Standard Deviation); unit: cm] | 171.5 (10.47) | 172.8 (10.39) | 171.6 (9.99) | 170.7 (11.16) | 173.4 (9.63) | 172.0 (10.27)
Weight [Mean (Standard Deviation); unit: kg] | 100.76 (25.675) | 108.52 (25.451) | 103.75 (27.027) | 96.43 (21.749) | 98.44 (22.844) | 101.58 (24.749)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 34.08 (6.993) | 36.53 (9.036) | 35.23 (8.655) | 33.10 (7.220) | 32.62 (6.609) | 34.31 (7.810)
Smoking History [Number; unit: participants]
  Never Smoked | 20 | 21 | 19 | 20 | 16 | 96
  Current Smoker | 2 | 3 | 4 | 5 | 5 | 19
  Ex-Smoker | 16 | 13 | 16 | 12 | 17 | 74
Alcohol Classification [Number; unit: participants]
  Never Drank | 8 | 14 | 14 | 19 | 20 | 75
  Current Drinker | 22 | 15 | 15 | 14 | 13 | 79
  Ex-Drinker | 8 | 8 | 10 | 4 | 5 | 35

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serum Urate <5.0 mg/dL at Month 3
Time Frame: Month 3
Population: Full Analysis Set (FAS) included all participants who were randomized and received at least 1 dose of double-blind study medication. Participants who discontinued double-blind study drug prior to the Month 3 visit were considered treatment failures, i.e. to have serum urate ≥ 5.0 mg/dL.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg
Number analyzed (Participants) | 38 | 37 | 39 | 37 | 38
percentage of participants | 0 | 13.5 | 35.9 | 40.5 | 44.7
Statistical Analysis 1: Comparison: Placebo vs Febuxostat XR 40 mg; Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 35.9, 95% CI 2-sided [20.8 to 51.0]
Statistical Analysis 2: Comparison: Placebo vs Febuxostat XR 80 mg; Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 44.7, 95% CI 2-sided [28.9 to 60.5]
Statistical Analysis 3: Comparison: Febuxostat IR 40 mg vs Febuxostat XR 40 mg; Test type: Superiority or Other; p = 0.034, Fisher Exact; Difference in Proportions = 22.4, 95% CI 2-sided [3.7 to 41.0]
Statistical Analysis 4: Comparison: Febuxostat IR 80 mg vs Febuxostat XR 80 mg; Test type: Superiority or Other; p = 0.817, Fisher Exact; Difference in Proportions = 4.2, 95% CI 2-sided [-18.2 to 26.6]

2. Secondary Outcome: Percentage of Participants With at Least One Gout Flare Requiring Treatment
Description: A participant was considered to have a gout flare if the following criteria were met:
  Participant-reported acute particular pain typical of a gout attack that was deemed by participant and/or investigator to require treatment and was treated with colchicine, nonsteroidal anti-inflammatory drugs (NSAIDs) or steroids, Participant experienced at least 3 or more of: 1) Joint swelling, 2) Redness, 3) Tenderness, 4) Pain, Participant experienced at least one or more of: 1) Rapid onset of pain, 2) Decreased range of motion, 3) Joint warmth, 4) Other symptoms similar to a prior gout flare.
Time Frame: Baseline to Month 3
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg
Number analyzed (Participants) | 38 | 37 | 39 | 37 | 38
percentage of participants | 10.5 | 40.5 | 23.1 | 37.8 | 42.1
Statistical Analysis 1: Comparison: Placebo vs Febuxostat XR 40 mg; Test type: Superiority or Other; p = 0.224, Fisher Exact; Difference in Proportions = 12.6, 95% CI 2-sided [-3.9 to 29.0]
Statistical Analysis 2: Comparison: Placebo vs Febuxostat XR 80 mg; Test type: Superiority or Other; p = 0.004, Fisher Exact; Difference in Proportions = 31.6, 95% CI 2-sided [13.1 to 50.1]
Statistical Analysis 3: Comparison: Febuxostat IR 40 mg vs Febuxostat XR 40 mg; Test type: Superiority or Other; p = 0.139, Fisher Exact; Difference in Proportions = -17.5, 95% CI 2-sided [-38.1 to 3.2]
Statistical Analysis 4: Comparison: Febuxostat IR 80 mg vs Febuxostat XR 80 mg; Test type: Superiority or Other; p = 0.815, Fisher Exact; Difference in Proportions = 4.3, 95% CI 2-sided [-17.9 to 26.4]

3. Secondary Outcome: Percentage of Participants With Serum Urate <6.0 mg/dL at Month 3
Time Frame: Month 3
Population: FAS included all participants who were randomized and received at least 1 dose of double-blind study medication. Participants who discontinued double-blind study drug prior to the Month 3 visit were considered treatment failures, i.e. to have serum urate ≥ 5.0 mg/dL.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg
Number analyzed (Participants) | 38 | 37 | 39 | 37 | 38
percentage of participants | 0 | 32.4 | 53.8 | 59.5 | 55.3
Statistical Analysis 1: Comparison: Placebo vs Febuxostat XR 40 mg; Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 53.8, 95% CI 2-sided [38.2 to 69.5]
Statistical Analysis 2: Comparison: Placebo vs Febuxostat XR 80 mg; Test type: Superiority or Other; p < 0.001, Fisher Exact; Difference in Proportions = 55.3, 95% CI 2-sided [39.5 to 71.1]
Statistical Analysis 3: Comparison: Febuxostat IR 40 mg vs Febuxostat XR 40 mg; Test type: Superiority or Other; p = 0.069, Fisher Exact; Difference in Proportions = 21.4, 95% CI 2-sided [-0.3 to 43.1]
Statistical Analysis 4: Comparison: Febuxostat IR 80 mg vs Febuxostat XR 80 mg; Test type: Superiority or Other; p = 0.817, Fisher Exact; Difference in Proportions = -4.2, 95% CI 2-sided [-26.6 to 18.2]

ADVERSE EVENTS:
Time Frame: First dose of double-blind study drug to 30 days past last dose of double-blind study drug (Up to 4 Months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Febuxostat IR 40 mg | Febuxostat XR 40 mg | Febuxostat IR 80 mg | Febuxostat XR 80 mg
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/37 | 1/39 | 0/37 | 4/38
Other Adverse Events (participants affected / at risk) | 3/38 | 5/37 | 4/39 | 1/37 | 3/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Febuxostat IR 40 mg (N=37) | Febuxostat XR 40 mg (N=39) | Febuxostat IR 80 mg (N=37) | Febuxostat XR 80 mg (N=38)
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Sinus node dusfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with febuxostat XR 80 mg and is not related.
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=38) | Febuxostat IR 40 mg (N=37) | Febuxostat XR 40 mg (N=39) | Febuxostat IR 80 mg (N=37) | Febuxostat XR 80 mg (N=38)
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.